CLINICAL TRIAL: NCT01936636
Title: Rapid Evaluation of Lifestyle, Independence, and Elimination of Breakthrough Cancer Pain With Freedom From Oral Discomfort Through the Use of Abstral® (Fentanyl) Sublingual Tablets
Brief Title: Observational Registry Study of Quality of Life When Treating BTcP With Abstral
Acronym: RELIEF
Status: Completed | Type: Observational
Sponsor: Galena Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RELIEF
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Quality of Life; Breakthrough Cancer Pain
Keywords: Breakthrough cancer pain; diary; quality of life; Abstral; BTcP
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients treated for BTcP: All patients 18 years of age and older with breakthrough cancer pain (BTcP) who are registered in the Transmucosal Immediate Release Fentanyl (TIRF) Risk Evaluation and Mitigation Strategy (REMS) Access program and receiving Abstral® under the direction of a TIRF REMS Access program-registered physician are eligible for the study.
  Patients or their proxy with a witness must be able to sign written informed consent to participate in the study; and the patient may also use a proxy caregiver to assist in the completion of the study questionnaires.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl

SUMMARY:
This Observational Registry study is designed to collect self-reported Transmucosal Immediate Release Fentanyl (TIRF) Risk Evaluation and Mitigation Strategy (REMS) Access program-enrolled patient experience with breakthrough cancer pain (BTcP) as a result of treatment with Abstral® through the use of Quality of Life and pain measurement tools administered via questionnaire.

DETAILED DESCRIPTION:
This is a post-marketing, single arm, open label multicenter trial to assess Abstral (fentanyl) Sublingual Tablets for breakthrough cancer pain (BTcP) in opioid-tolerant cancer patients.

* Prior to study enrollment, patient enrollment in the TIRF REMS Access program must be confirmed.
* Eligible patients will sign written informed consent. Patients or their proxy with a witness must be able to sign written informed consent to participate in the study; and the patient may use a proxy caregiver to assist in the completion of the study questionnaires.
* Day 0, study site must enroll patient by completing a patient demographic profile (de-identified).
* Day 0, patient will be instructed how to use the questionnaires.
* Day 0, patient will complete the baseline questionnaire before leaving the physician office.
* On study Days 14, 21, and 28 (±3 days) patient questionnaire will be completed by patient (or caregiver proxy) via secure online data entry portal.
* For patients completing paper questionnaires, within 1 month of day 28, patient will return completed questionnaires via mail, fax or hand carried to the study site coordinator for processing.
* Patient will be considered to have completed the study successfully once all completed questionnaires have been received by the CRO within appropriate time limits.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older with breakthrough cancer pain who are registered in the Transmucosal Immediate Release Fentanyl (TIRF) Risk Evaluation and Mitigation Strategy (REMS) Access program and receiving Abstral® under the direction of a TIRF REMS Access program-registered physician are eligible for the study.

Patients or their proxy with a witness must be able to sign written informed consent to participate in the study; and the patient may also use a proxy caregiver to assist in the completion of the study questionnaires.

Exclusion Criteria:

* No patient can be enrolled who has not been prescribed Abstral for BTcP in compliance with Transmucosal Immediate Release Fentanyl (TIRF) Risk Evaluation and Mitigation Strategy (REMS) Access program guidelines.

No patient may be enrolled who has a contraindication to receiving Abstral or who is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational Registry study is designed to collect self-reported TIRF REMS Access program-enrolled patient experience with breakthrough cancer pain (BTcP) as a result of treatment with Abstral® through the use of Quality of Life and pain measurement tools administered via questionnaire.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | One month
  Primary:
  To compare self reported TIRF REMS Access-enrolled patient experience with BTcP at baseline (before using Abstral) to their experience after reaching a maintenance dose of Abstral
  * Characterize the effectiveness of treatment with Abstral in select pain and quality-of-life (QoL) domains
  * Abstral impact on pain interference with daily activities, somnolence, and oral health

SECONDARY OUTCOMES:
Rapidity of BTcP | one month
  Trends in improvement or deterioration in these values during treatment and across the dosage groups will be described.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Physicians Pain Specialists of Alabama, P.C., Mobile, Alabama
  - Pain Centers Nationwide, Peoria, Arizona
  - Valley Pain Consultants, Scottsdale, Arizona
  - Coastal Pain Research, Carlsbad, California
  - Navajo Road Pain Management Center, El Cajon, California
  - California Cancer Associates for Research and Excellence, Inc., Fresno, California
  - Interventional Pain Management, Irvine, California
  - Alexander Ford, MD, Los Angeles, California
  - Cancer Care Institute, Los Angeles, California
  - Pete J. Ruane, MD, Inc., Los Angeles, California
  - Pain Institute of Santa Monica, Santa Monica, California
  - Randy Scharlach, MD, Woodland Hills, California
  - Red Rocks Center for Rehabilitation, Golden, Colorado
  - Western Connecticut Health Network, Danbury Hospital, Danbury, Connecticut
  - Pain Management Associates of CT, PC, Stamford, Connecticut
  - Florida Cancer Care, Plantation, Florida
  - Interventional Spine and Pain Management, Atlanta, Georgia
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Pain Management Institute, Overland Park, Kansas
  - Physiatry Consultants, Bay City, Michigan
  - Michigan Interventional Pain Center, Brownstown, Michigan
  - Glenn Saperstein, D.O., LLC, Saginaw, Michigan
  - Advanced Physical Medicine, Saint Clair Shores, Michigan
  - Michigan Spine & Pain, West Bloomfield, Michigan
  - Fountain Medical Group, New York, New York
  - Upper East Side Pain Medicine, P.C., New York, New York
  - Comprehensive Pain Management, Syosset, New York
  - APWI, Williamsville, New York
  - Akron General Medical Center, Akron, Ohio
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - J. Fred Stoner, MD, New Castle, Pennsylvania
  - Progressive Pain Solutions, Wind Gap, Pennsylvania
  - Jerrold Rosenberg, MD, Providence, Rhode Island
  - The West Clinic Comprehensive Breast Center, Germantown, Tennessee
  - PRIDE, Dallas, Texas
  - Columbia Basin Hematology & Oncology, Kennewick, Washington